CLINICAL TRIAL: NCT07071077
Title: Examining the Feasibility of Implementing a Hypertension Storytelling Intervention Among African Americans With Hypertension
Brief Title: Examining the Feasibility of Implementing a Hypertension Storytelling Intervention Among African Americans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Yendelela Cuffee, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2034724-5; 5K01HL166372-02 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Medication Adherence; Lifestyle Intervention; Behavioral Change
MeSH Terms: conditions — Hypertension; Medication Adherence | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention)
- Storytelling (Web-based Storytelling) (Experimental)
  Interventions: Behavioral: Web-Based Storytelling Intervention
- Storytelling Plus (Group-based Storytelling) (Experimental)
  Interventions: Behavioral: Group-Based Storytelling Plus Intervention

INTERVENTIONS:
Behavioral: Web-Based Storytelling Intervention — The Web-based storytelling group will access stories and educational materials on the study website.
  Arms: Storytelling (Web-based Storytelling)
Behavioral: Group-Based Storytelling Plus Intervention — The storytelling plus group will watch the stories in a group setting, share their experiences and have educational sessions led by a health coach.
  Arms: Storytelling Plus (Group-based Storytelling)

SUMMARY:
The purpose of this study is to assess if storytelling is an effective approach for promoting lifestyle and behavioral change among individuals managing hypertension and to determine if storytelling interventions can help to reduce blood pressure and improve medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black
* Diagnosed with Hypertension
* Prescribed medication for hypertension

Exclusion Criteria:

* Cognitive limitations that limit the ability to provide informed consent
* Pregnancy
* Unable to speak or read English
* Planning to relocate during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood Pressure | 6 months
  Blood pressure will be measured three times using a manual blood pressure monitor.
Adherence to Antihypertensive Medications (daily usage) | 6 months
  Medication adherence will be measured using Medication Electronic Measuring System (MEMS) caps
Adherence to Antihypertensive Medications (self reported) | 6 months
  Medication adherence will be measure through participant self report Domains of Subjective Extent of Nonadherence scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided